CLINICAL TRIAL: NCT05893615
Title: Effects of Cognitive Behavior Therapy on Anxiety, Depression, Illness Perception, and Quality of Life in Paroxysmal Atrial Fibrillation Patients
Brief Title: Effects of Cognitive Behavior Therapy on Quality of Life in Paroxysmal Atrial Fibrillation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Qu Shan, Head of the Department of Medical Psychology, Peking University People's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AF-CBT-HRQoL2020
Record Dates: First submitted 2023-05-26; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: CBT
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT group (Active Comparator): Patients in the CBT intervention group, who received CBT focused on anxiety symptoms in addition to their usual treatment, including 10 one-hour sessions spread over 10 weeks, and weekly homework guided by the therapist.
  Interventions: Behavioral: Cognitive Behaviour Therapy
- Treatment as usual (TAU) group (No Intervention): Patients in TAU group received optimal medical care according to the current clinical guidelines. Patients in the TAU group did not receive any psychotherapy.

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy — The CBT module was adjusted as follows: (1) Health education about paroxysmal atrial fibrillation; (2) Self-awareness training; (3) Exposure training; (4) Habitual reversal training；(5) Correcting cognitive distortion; (6) Behavioral activation (7) Specific training for anxiety; (8) Practice and feedback; (9) Relapse prevention; (10) Review.
  Arms: CBT group

SUMMARY:
Health-Related Quality of Life (HRQoL) was commonly impaired in atrial fibrillation patients. Depression, anxiety, and illness perception are psychological correlates of HRQoL. Our previous study had shown good effects of CBT on the quality of life in AF patients. This study aimed to establish the long-term efficacy of CBT on both psychological distress and HRQoL. Method: The study was a prospective, open study, pseudo-randomization with a pretest-posttest design and a 6-month follow-up. A total of 102 patients with paroxysmal AF were enrolled, and 90 patients were assigned (1:1) to 10 weeks of CBT focused on anxiety symptoms or to treat as usual in the end. Item Short Form Health Survey (SF-12), GAD-7, PHQ-9, University of Toronto Atrial Fibrillation (AFSS), and Brief Illness Perception Questionnaire (BIPQ) were measured as outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for participation were: (a) age 18-75 years; (b) AF diagnosis, based on a 12-lead ECG and cardiologist-led examination following the 2016 ESC Guidelines for the Management of Atrial Fibrillation5 and (c) paroxysmal AF diagnosis given by a cardiologist according to the conversion back to the normal sinus rhythm occurs spontaneously within a week 18. (d) ability to read and write in Chinese.

Exclusion Criteria:

* (a) severe complications such as unstable coronary artery disease, heart failure with severe systolic dysfunction(ejection fraction≤35%); (b)AF soon after thoracic surgery; (c) malignant disease with a 1-year survival rate or a terminal illness diagnosis; (d) a diagnosed psychiatric condition that interfered with participation (including severe depression, bipolar disorder, psychotic illness of any type, dementia, acute suicidality, severe personality disorder);(e) regular psychological therapy with a mental health condition; (f) participation in another study; (g) cognitive impairment interfering with their ability to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline score of The 12-item Health Survey Short Form (SF-12) at 10 weeks and 6 months | Both groups were assessed the SF-12 three times, respectively at baseline, 10 weeks later and 6 month later
  SF-12 is a 12-item, multipurpose short-form survey that is used to measure generic HRQoL (derived from the SF-36). The findings are weighted and summed to produce interpretable scales for a participant's physical and mental well-being. SF-12 is divided into two domains: the physical component summary (PCS) and the mental component summary (MCS). Each domain scores from 0 to 100, with higher scores indicating a better health status

SECONDARY OUTCOMES:
Brief Illness Perception Questionnaire (BIPQ) | Both groups were assessed the BIPQ three times, respectively at baseline, 10 weeks later and 6 month later
  The Brief Illness Perception Questionnaire (BIPQ) is a nine-item questionnaire that assesses how people feel about illnesses across nine categories. The individual nine domain scores were added together to create a composite BIPQ score. A higher BIPQ score suggests that the psychological burden of illness is greater (range: 0-80). The BIPQ assesses the following illness perception domains: identity (symptoms experienced); timeline-acute/chronic (perception of the length of disease); consequences (effect of disease on one's life); personal control (control over disease); treatment control (perception of treatment impact); emotional representations (emotional effect of the disease); illness coherence (understanding of disease); illness concern (concern about the disease); and cause (perceived cause of disease). The cause item is an open-ended question that asks patients to rank the top three factors they believe caused their disease
University of Toronto Atrial Fibrillation Severity Scale (AFSS) | Both groups were assessed the AFSS symptoms subscale three times, respectively at baseline, 10 weeks later and 6 month later
  University of Toronto Atrial Fibrillation Severity Scale (AFSS)-a 14-item disease-specific scale consisting of three parts. Part 1 measures patients with atrial fibrillation overall life satisfaction and frequency, duration of atrial fibrillation attacks, and severity; Part 2 measures patient utilization rates; Part 3 is divided into symptom subscales, including 7 common symptoms of atrial fibrillation (heart palpitations, dyspnea at rest, dyspnea with activity, exercise intolerance, vertigo, fatigue at rest, and chest pain) and the corresponding frequency of attacks. In this study, the symptom part was selected as the AF symptoms measurement.
The Generalized Anxiety Disorder Questionnaire (GAD-7) | Both groups were assessed the GAD-7 three times, respectively at baseline, 10 weeks later and 6 month later
  The Generalized Anxiety Disorder Questionnaire (GAD- 7) is a 7-item measure of anxiety symptoms, using a four-point Likert-type scale. The GAD-7 asks how often people have suffered from the seven core symptoms of GAD within the last two weeks with the response options being 'not at all', 'on some days', 'on more than half of the days', and 'almost every day' (scored 0-3, with a total score ranging from 0 to 21). A sum score of≥10 indicates clinically relevant anxiety.
The Patient Health Questionnaire-9 (PHQ-9) | Both groups were assessed the PHQ-9 three times, respectively at baseline, 10 weeks later and 6 month later
  The Patient Health Questionnaire-9 (PHQ-9) is a nine-item tool used to measure the severity of depression over the previous 2 weeks (range 0-27). he PHQ-9 was chosen above other depression screening measures because it is easy to administer and outperforms the structured clinical interview for the Diagnostic and Statistical Manual of Mental Disorders-IV as the standard criterion.

CONTACTS AND LOCATIONS:
Overall Officials: Qu Shan, Principal Investigator — Peking University People's Hospital
Locations (1):
- Minjie Zheng, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No